CLINICAL TRIAL: NCT02216513
Title: Deferoxamine: An Emerging Therapy to Prevent Delayed Cerebral Ischemia After Subarachnoid Hemorrhage
Brief Title: Deferoxamine to Prevent Delayed Cerebral Ischemia After Subarachnoid Hemorrhage
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Principle Investigator is moving to another institution and plans to restart this proctocol in the new location.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Dr. Jeffrey Thomas Stroke Shield Foundation (Unknown)
Responsible Party: Principal Investigator, Farzaneh Sorond, BWPO Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014P001400
Record Dates: First submitted 2014-08-06; First posted 2014-08-15 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Subarachnoid Hemorrhage
Keywords: subarachnoid hemorrhage; SAH; DFO; cerebral autoregulation; delayed cerebral ischemia
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Deferoxamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desferrioxamine (DFO) (Active Comparator): DFO (20mg/kg/hr) in normal saline IV for 4 hours for 5 consecutive days
  Interventions: Drug: desferrioxamine (DFO)
- placebo (Placebo Comparator): normal saline IV for 4 hours for 5 consecutive days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: desferrioxamine (DFO) — DFO (20mg/kg/hr) in normal saline for 4 hours for 5 consecutive days
  Other Names: deferoxamine, desferal, DFO, deferoxamine mesylate
  Arms: Desferrioxamine (DFO)
Drug: placebo — normal saline IV for 4 hours for 5 consecutive days
  Other Names: normal saline NS
  Arms: placebo

SUMMARY:
The investigators will test the central hypothesis that DFO treatment after SAH may improve cerebrovascular regulation, mitigate ischemic neural injury, and serve as an effective neuroprotectant against delayed ischemic injury after SAH.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of spontaneous SAH
* impaired cerebral autoregulation on day 2-4 post SAH

Exclusion Criteria:

* traumatic SAH
* other central neurological disorders such as tumors, known prior stroke, hemorrhage or vascular malformations
* pregnancy
* severe renal disease or anuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
delayed cerebral ischemia (DCI) | 6 weeks post hemorrhage
  DCI will be defined radiographically as any cerebral infarct on the latest CT scan that was seen within 6 weeks after SAH or before discharge or death, that was not present on admission scan or on the CT scan done within 24 to 48 hours after any aneurysmal treatment procedures. All head CT scans will be reviewed for DCI ascertainment by neuroradiologists blinded to the clinical and TCD data using the standardized protocol.

SECONDARY OUTCOMES:
Clinical outcome at discharge | patient's discharge date, which averages 3-4 weeks post hemorrhage
  Clinical outcome at discharge will be assessed using modified Rankin Scale (mRS) as a global functional status. The modified Rankin scale evaluates global disability and handicap; scores range from 0 (no symptoms or disability) to 6 (death). Good mRS will be defined as score of ≤ 2.

OTHER OUTCOMES:
Cerebrovascular function (i.e., cerebral autoregulation) | 5 days after initiation of study drug
  Spectral analysis of the relationship between arterial pressure and blood flow velocity in the bilateral middle cerebral arteries (measured via TCD). Autoregulation will be assessed from the phase and gain of the transfer function. Phase shift reflects the temporal difference between cerebral flow velocity fluctuations with respect to arterial pressure fluctuations. When the fluctuations of both flow and pressure are almost synchronous, the phase shift approaches zero, reflecting impaired cerebral autoregulation. Transfer function gain reflects the magnitude of transmission of arterial pressure fluctuations to cerebral blood flow velocity fluctuations. Lower gain, particularly in the low frequency (< 0.1 Hz) range, is reflective of more effective cerebral autoregulation. Coherence reflects the degree of linear dependence between pressure and flow fluctuations. Thus, it provides a measure of validity of the metrics (gain and phase) derived from the linear transfer function.

CONTACTS AND LOCATIONS:
Overall Officials: Farzaneh A Sorond, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Van der Loo LE, Aquarius R, Teernstra O, Klijn K, Menovsky T, van Dijk JMC, Bartels R, Boogaarts HD. Iron chelators for acute stroke. Cochrane Database Syst Rev. 2020 Nov 24;11(11):CD009280. doi: 10.1002/14651858.CD009280.pub3. PMID 33236783